CLINICAL TRIAL: NCT00006496
Title: Molecular Epidemiology of Acute Respiratory Distress Syndrome
Brief Title: Molecular Epidemiology of Acute Respiratory Distress Syndrome (ARDS)
Status: Active, not recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, David Christopher Christiani, Professor of Medicine, Massachusetts General Hospital
Other Study IDs: 937; R01HL060710 (NIH)
Record Dates: First submitted 2000-11-16; First posted 2000-11-17 (Estimated); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Acute Respiratory Distress Syndrome; Lung Diseases
MeSH Terms: conditions — Respiratory Distress Syndrome; Lung Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood will be collected for DNA extraction and plasma cytokine measurements
Oversight: Data Monitoring Committee: No

SUMMARY:
To examine the possible relationship between genetic factors and the acute respiratory distress syndrome (ARDS).

DETAILED DESCRIPTION:
BACKGROUND:

The acute respiratory distress syndrome (ARDS) remains a major cause of morbidity and mortality around the world. In the United States alone there are 150,000 cases per year. Although there have been significant scientific advances in understanding the clinical and pathophysical aspects of the syndrome, there is as yet no specific therapy for ARDS. Moreover, although major risk factors for the development of ARDS include sepsis, aspiration, and multiple trauma, only a minority of patients with these risk factors develop ARDS. Individual differences in susceptibility to chronic disease have been a subject of active molecular epidemiologic investigations for the past decade. In particular, risk factors for cancer conferred by heritable polymorphisms and various metabolic functions have been reported. More recently, a polymorphism of endothelial nitrate oxide synthase has been associated with an increased susceptibility to coronary-artery disease, and polymorphisms in GSTM1 have been associated with an increased risk of developing asbestosis. A recent study of tumor necrosis factor (TNF) polymorphisms has been associated with poor outcome in ARDS.

DESIGN NARRATIVE:

The case-control study examined the association between specific polymorphisms in several genes coding for specific inflammatory responses and for surfactant protein and their potential association with increased susceptibility to ARDS. The first objective was to assess the role of candidate-gene polymorphisms as risk factors for ARDS in a case-control study. The second objective was to assess the relationship between genotype and phenotype for candidate markers in cases and controls. The third objective was to assess the role of these polymorphisms in clinical outcome (survival, recovery) using patients from both the proposed case-control study and the multicenter case series and clinical trial sponsored by the NHLBI ARDS network. By combining both a large case-control study and case series from the network, the study had the advantages of sufficient case ascertainment, statistical power, diagnostic standardization, uniform outcome criteria and study efficiency. Overall, the results of this study should provide new insights into the epidemiology of ARDS and allow for possible preventive strategies as well as possible modifications of therapeutic interventions for the Network Phase III trials.

The investigators test the hypothesis that there is an increased risk of ARDS in patients with heritable traits relating to inflammatory cytokines and surfactant. They are examining risk and prognosis, and examining case and control genetics in relation to cytokine levels. They also plan to do a case-series analysis from a separate study of the ARDS network. They will examine TNF alpha and beta, interleukin-1 receptor antagonist, surfactant protein B and interleukin-10 (IL-10).

ELIGIBILITY:
Eligibility Criteria:

All those with risk factors for ARDS - eg, pneumonia, trauma, sepsis.

Vulnerable populations (incarcerated, pregnant, etc.) will be excluded from enrollment. The following medical conditions will also exclude from study:

1. immunocompromised patients
2. patients with chronic lung disease that may appear like ARDS
3. pulmonary vasculitis patients
4. patients with diffuse alveolar hemorrhage
5. patients treated with immune-modulating agents within 3 weeks of admission
6. patients unable to intubate because of DNI order or patient is placed on comfort measures only

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to ICU with risk factors for ARDS
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2000-02; Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Risk of ARDS | From admission to ICU

SECONDARY OUTCOMES:
Mortality | From admission to ICU to 60 days

OTHER OUTCOMES:
Multi-organ Failure | From admission to ICU

CONTACTS AND LOCATIONS:
Overall Officials: David Christiani, MD, Principal Investigator — Harvard University School of Public Health
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gong MN, Wei Z, Xu LL, Miller DP, Thompson BT, Christiani DC. Polymorphism in the surfactant protein-B gene, gender, and the risk of direct pulmonary injury and ARDS. Chest. 2004 Jan;125(1):203-11. doi: 10.1378/chest.125.1.203. PMID 14718442
- [Background] Gong MN, Thompson BT, Williams P, Pothier L, Boyce PD, Christiani DC. Clinical predictors of and mortality in acute respiratory distress syndrome: potential role of red cell transfusion. Crit Care Med. 2005 Jun;33(6):1191-8. doi: 10.1097/01.ccm.0000165566.82925.14. PMID 15942330